CLINICAL TRIAL: NCT03858699
Title: Brain Vital Signs M-Score: Point-of-care Monitoring for Motor Recovery After Stroke
Status: Terminated | Type: Observational
Why Stopped: low recruitment
Sponsor: HealthTech Connex Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HTC_MScore_001
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with stroke: Participants in sub-acute and chronic phases post-stroke (>1 month post-stroke) will be recruited for participation in this study.
  Interventions: Other: Recording of electroencephalographic (EEG) data
- Adult control participants: Even age distributions will be recruited in the adult control group, stratified under 40 years old and over 40 years old.
  Interventions: Other: Recording of electroencephalographic (EEG) data

INTERVENTIONS:
Other: Recording of electroencephalographic (EEG) data — Non-invasive brain activity will be measured with electroencephalography (EEG). EEG uses scalp sensors to monitor the brain's electrical activity. EEG sensors are placed on the scalp and passively record neural activity with high time resolution.

SUMMARY:
The purpose of this study is to investigate brain signals relating to motor function, using electroencephalography (EEG) technology. The aims of the study can be separated into 3 specific study objectives:

1. Record EEG data from control participants and individuals with stroke during basic motor tasks and build a database of EEG signals to enable analysis of motor control.
2. Apply signal processing algorithms to extract EEG features related to motor control.
3. Develop a framework/the motor score (M-Score) that uses the EEG signals, in combination with machine learning approaches, to quantify motor control ability.

ELIGIBILITY:
Inclusion Criteria:

* Age requirements:

  * Younger adult control participants (19-40 years old)
  * Older adult control participants (41-80 years old)
  * Individuals with stroke (19-80 years old)
* Capacity to follow single stage commands
* Stroke specific inclusion criteria

  * Upper-limb disability as a result of a stroke (>1 month ago)

Exclusion Criteria:

* Cognitive difficulties that undermine ability to give informed consent (Montreal Cognitive Assessment (MoCA) score below 23).
* Severe paralysis such that the participant cannot perform simple movements (such as finger tapping, clicking a mouse, etc.)
* History of head trauma, a major psychiatric diagnosis, neurodegenerative disorder or substance abuse

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Number of Participants: Up to 30 healthy participants and 30 individuals with stroke.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Resting state EEG measures | 1 day
  EEG uses scalp sensors to monitor the brain's electrical activity. EEG sensors are placed on the scalp and passively record neural activity with high time resolution. The principal recording system for this study will be a 32-channel g.Nautilus EEG system (g.tec medical engineering). Secondary recording systems may be used: 8-channel g.Nautilus EEG system (g.tec medical engineering) and 64-channel, high-density BrainAmp EEG system (BrainProducts).Participants will be seated while wearing the EEG cap and asked to sit quietly with either eyes open (with a fixation dot or cross to reduce eye movements) or eyes closed. Resting state recordings will be approximately 5-10 minutes in length.
Motor task EEG measures | 1 day
  While completing EEG scans, participants will be asked to execute simple motor movements. . Study will focus on finger tapping task (with mouse-like button for recording movement timing). Participants will be asked to complete self-paced movements with approximately 10-15 second inter-trial spacing. Recording will occur in two-minute intervals, followed by a rest period, repeated until approximately 40 trials have been collected. Other motor movements, such as flexion of the upper limbs or flexion of the lower limbs, may also be considered. During EEG recordings changes in motor oscillations (alpha, beta, & gamma range) will be analyzed. During EMG recordings, muscle tonicity/spasticity and functional firing patterns will be analyzed.
Imagery task EEG measures | 1 day
  During EEG recording participants could be asked to engage in mental imagery of motor movements stated above. Here, potential changes in oscillatory patterns in the motor cortex will be measured and detected.

SECONDARY OUTCOMES:
Wolf Motor Function Test | 1 day
  The Wolf Motor Function Test (WMFT) quantifies upper extremity motor ability using timed functional tasks.
Fugl-Meyer Assessment | 1 day
  The Fugl-Meyer Assessment (FMA) is a performance-based impairment index designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia.
Box-and-Block Test | 1 day
  This test is used to quantify the gross manual dexterity of each hand and arm.
Nine-Hole Peg Test | 1 day
  This test is used to quantify the fine manual dexterity of each hand and arm.

CONTACTS AND LOCATIONS:
Locations (1):
- HealthTech Connex Centre for Neurology Studies, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No